CLINICAL TRIAL: NCT06199882
Title: A Single-arm, Open, Single-center Phase II Clinical Study on the Efficacy and Safety of SBRT Sequential Surufatinib Combined With Immunotherapy for Locally Unresectable or Recurrent Biliary Tract Cancer After First Surgery
Brief Title: SBRT Sequential Surufatinib Combined With Immunotherapy for Biliary Tract Carcinoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient recruitment difficulties
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Liu luying, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-383
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT Sequential Surufatinib Combined With Immunotherapy (Experimental): SBRT :
  Bioequivalent total dose > 75Gy, completed within 2 weeks (once daily, 5 times a week).
  Drug treatment (every 3 weeks is a treatment cycle) :
  1) Surufatinib: 200 mg, po, qd, taken continuously; 2) Carrelizumab: 200 mg/ time, intravenous drip on the first day of each cycle.
  Interventions: Drug: SBRT Sequential Surufatinib Combined With Immunotherapy

INTERVENTIONS:
Drug: SBRT Sequential Surufatinib Combined With Immunotherapy — 1. SBRT :
     Bioequivalent total dose > 75Gy, completed within 2 weeks (once daily, 5 times a week).
  2. Drug treatment (every 3 weeks is a treatment cycle) :
  1) Surufatinib: 200 mg, po, qd, taken continuously; 2) Carrelizumab: 200 mg/ time, intravenous drip on the first day of each cycle.
  Other Names: SBRT--Surufatinib+Carrelizumab

SUMMARY:
This is a single-arm, open, single-center Phase II clinical study to observe and evaluate the efficacy and safety of SBRT sequential surufatinib combined with immunotherapy in patients with locally unresectable or recurrent biliary tract cancer after the first surgery.

DETAILED DESCRIPTION:
This is a single-arm, open, single-center Phase II clinical study to observe and evaluate the efficacy and safety of SBRT sequential surufatinib combined with immunotherapy in patients with locally unresectable or recurrent biliary tract cancer after the first surgery.The study was divided into three stages: screening period, treatment period and follow-up period. During treatment, imaging methods were used to evaluate tumor status every 6 weeks (±7 days) until disease progression (PD, RECIST 1.1) or death (during treatment) or toxicity became intolerable, and tumor treatment and survival status after disease progression were recorded. Safety outcome measures included AE, changes in laboratory test values, vital signs and electrocardiogram changes.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in this study, patients must meet all of the following criteria:

  1. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up;
  2. Age 18-75 years old (including 18 and 75 years old), gender is not limited;
  3. Patients with unresectable or untreated recurrent BTC confirmed by histopathology or cytology (including intrahepatic, extrahepatic, and gallbladder cancers);
  4. Have not received any anti-tumor therapy before;
  5. Have at least one measurable lesion (according to RECIST 1.1 standards); Magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement were used to accurately measure the diameter ≥10mm, and conventional CT scan was used to measure the diameter at least 20mm.
  6. Normal liver volume (total liver volume minus tumor GTV volume) exceeds 1000cc;
  7. The maximum diameter of the tumor is less than 10cm, allowing up to 3 satellite foci. Satellite foci were defined as being less than 2cm and within 1cm of the gross tumor.
  8. No serious organic diseases of heart, lung, brain and other organs;
  9. The main organs and bone marrow functions are basically normal:

  <!-- -->

  1. Blood routine: white blood cells ≥ 4.0 x 10^9/L, neutrophils ≥ 1.5 x 10^9/L, platelets ≥ 80 x 10^9/L, hemoglobin ≥ 90g/L;
  2. International Standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5× upper limit of normal (ULN);
  3. Liver function: serum total bilirubin ≤ 1.5 x ULN, ALT/AST ≤ 3 x ULN, serum total bilirubin ≤ 1.5 x ULN after internal/external drainage of obstructive jaundice;
  4. Renal function: serum creatinine ≤ 1.5x ULN, creatinine clearance (CCr) ≥ 50mL/min;
  5. Normal cardiac function with left ventricular ejection fraction (LVEF)≥50% as measured by two-dimensional echocardiography; Fertile male or female patients volunteered to use effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, and Iuds, during the study period and within 6 months of the last study medication. All female patients will be considered fertile unless the woman has undergone natural menopause, artificial menopause or sterilization.

Exclusion Criteria:

* The study proposal shall be excluded if any of the following criteria are met:

  1. Have received any antitumor therapy in the past (except simple surgical resection);
  2. The tumor directly invades the stomach, small intestine or colon;
  3. The maximum diameter of the lesion exceeds 10cm, or the satellite lesion does not meet the above definition criteria;
  4. Have had other malignancies within the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
  5. There are extra-hepatic metastases (excluding local regional lymph nodes);
  6. Normal liver volume is less than 1000cc;
  7. The patient currently has hypertension that cannot be controlled by drugs, as follows: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
  8. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume >1.0g;
  9. Patients whose tumors are judged by the investigators to be at high risk of invading vital blood vessels and causing fatal massive bleeding during the follow-up study;
  10. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months> 30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks > 5 mL fresh blood); Patients with a history of hereditary or acquired bleeding or coagulation disorders have clinically significant bleeding symptoms or definite bleeding tendencies within 3 months, such as gastrointestinal bleeding and hemorrhagic gastric ulcers;
  11. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure >Level 2; Ventricular arrhythmias requiring medical treatment; Electrocardiogram (ECG) showed QTC interval ≥480 ms.
  12. Active or uncontrolled severe infection (≥CTCAE grade 2 infection);
  13. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
  14. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, in which, in the investigator's judgment, there is reason to suspect that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or that would affect the interpretation of the study results or place the patient at high risk;
  15. Known human immunodeficiency virus (HIV) infection; Known history of clinically significant liver disease, including viral hepatitis [Known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis];
  16. The presence of any active, known or suspected autoimmune disease (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, pituitaries, hyperthyroidism, etc.);
  17. Allergy or suspected allergy to the investigational drug or similar drugs; According to the investigators' judgment, the patients had other factors that might affect the study results or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, and family or social factors that would affect the safety of the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | up to 12 months
  The proportion of subjects in the analyzed population who developed complete response (CR) and partial response (PR) according to RECIST (version 1.1) criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause
Local control rate (LCR) | up to 12 months
  The percentage of confirmed cases with complete response (CR), partial response (PR), and stable disease (SD) in patients for whom efficacy could be evaluated
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)
Incidence of adverse events （AE） | Until the last medication for 30 days (±7 days) or before the start of other anti-tumor therapy (whichever occurs first)
  Categorized according to NCI Common Toxicity Criteria version 5.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular forma

CONTACTS AND LOCATIONS:
Overall Officials: Luying Liu, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Liu luying, Hangzhou, Zhejiang, China